CLINICAL TRIAL: NCT03787199
Title: Feasibility of the Overground Bodyweight Supporting Walking System Andago
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: Lions Club Zürich-Witikon (Unknown); Mäxi Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018-00412
Record Dates: First submitted 2018-04-23; First posted 2018-12-26 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Gait Disorders, Neurologic; Cerebral Palsy; Stroke; Traumatic Brain Injury; Child, Only; Gait Disorders in Children
Keywords: Andago; Feasibility; Pediatric Neurorehabilitation
MeSH Terms: conditions — Gait Disorders, Neurologic; Cerebral Palsy; Stroke; Brain Injuries, Traumatic | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Feasibility study, including a comparison between Andago and treadmill walking conditions (as we include a heterogeneous group of participants concerning age (children/adolescents), diagnosis, walking ability, etc., we include in this feasibility study 20 participants - rather than the usual 10).
  Patients participate in 3 appointments (planned within 10 days):
  Appointment 1 (60 min): patient characteristics, clinical tests (Selective Control Assessment of the Lower Extremity / Manual Muscle Testing / 10 meter walk test or 10MWT); practising on treadmill and in Andago; questions to participants
  Appointment 2 (45 min): determine accuracy of the unloading system; practicing on treadmill and in Andago; questions to participant
  Appointment 3 (60-90 min): 10MWT at onset and end; measurement of stride length, leg muscle EMG and joint kinematics during walking on treadmill with bodyweight unloading and walking overground with Andago with 3 levels of bodyweight unloading
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Andago (Experimental): Application of walking over-ground with body-weight support in the Andago
  Interventions: Device: Andago
- Treadmill (Active Comparator): Application of walking on a treadmill with body-weight support
  Interventions: Other: Treadmill

INTERVENTIONS:
Device: Andago — The Andago is a body-weight supporting device with which a patient can walk overground
  Arms: Andago
Other: Treadmill — Bodyweight supported treadmill walking
  Arms: Treadmill

SUMMARY:
The overall aim of this project is to investigate the clinical utility of the Andago System, a CE certified mobile bodyweight supporting walking robot, in children with neuromotor disorders. Clinical utility encompasses practicability, acceptability, appropriateness, and accessibility. In this study, the investigators would like to investigate several aspects of clinical utility that belong to the first three components.

DETAILED DESCRIPTION:
The specific aims of the current project are:

1. To investigate the practicability, the investigators plan to determine the accuracy of the weight-supporting system of the Andago and the time needed for donning and doffing. The investigators also evaluate the number of times that the device stops and the nature of these stops (due to errors, sitting of the patient, when preventing falls, or when the patient moves too fast).
2. To evaluate acceptability, the investigators plan to evaluate differences in motivation and measures reflecting safety (i.e. number of falls prevented) and subjective feeling of safety when patients walk with the Andago compared to walking with their usual walking aids.
3. To evaluate the appropriateness, the investigators are interested in differences between walking on a treadmill and walking overground with this device or changes that occur during walking overground when changing the level of BWS through the unloading system. Therapists should be aware of these differences to know what the advantage of such a system could be or how adjustments in settings influence the walking pattern. The investigators plan two investigations: (a) To determine differences in stride-to-stride variability, leg muscle activation, hip, knee and ankle joint kinematics and other gait parameters during walking in the Andago (overground) versus walking on a treadmill. (b) To determine differences in the same parameters when walking in the Andago with different levels of BWS. These levels are the minimal required level of BWS to walk without buckling the knees (ref BWS), ref BWS plus 15% and ref BWS plus 30%.

To investigate these aims, the patients will be asked to participate in 3 appointments, which should be scheduled within 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Neuromotor or orthopaedic disorders
* taller than 135 cm
* able to understand simple instructions
* able to walk 10 meters with or without walking aid
* maximal age of 18 years (a minimal age is not defined as according to the growth curve, children younger than 7-8 years cannot be included because of insufficient height)
* given informed consent.

Exclusion Criteria:

* not consolidated fractures or bone fragility of the lower extremities
* skin lesions in the harness' area which cannot be protected
* unstable hip, knee and/or ankle Joints
* reduced head control or inability to maintain an upright Position
* inability to communicate discomfort or pain
* surgery in the last 3 months
* newly implanted baclofen-pump (or children highly sensitive to it)
* implanted pacemakers
* passive knee extension deficit > 30°
* self-selected walking speed > 3.2 km/h.
* weight > 135 kg
* height > 2 m.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Stride to stride variability | Appointment 3 (between minute 25 and minute 55 )
  Variability in stride length recorded during at least 20 steps for each of the following conditions: Andago with reference bodyweight support; Andago with 15% more bodyweight support; Andago with 30% more bodyweight support; and treadmill condition with reference bodyweight support

SECONDARY OUTCOMES:
Leg muscle activity | Appointment 3 (between minute 25 and minute 55 )
  Amplitude of electromyographic recordings recorded during at least 20 steps for each of the following conditions: Andago with reference bodyweight support; Andago with 15% more bodyweight support; Andago with 30% more bodyweight support; and treadmill condition with reference bodyweight support
Leg joint angles | Appointment 3 (between minute 25 and minute 55)
  Joint angles recorded with electrogoniometers during at least 20 steps for each of the following conditions: Andago with reference bodyweight support; Andago with 15% more bodyweight support; Andago with 30% more bodyweight support; and treadmill condition with reference bodyweight support

OTHER OUTCOMES:
Bodyweight unloading [kg] | Data are obtained during Appointment 2 (between minute 1 and minute 10)
  Comparison of bodyweight unloading according to Andago device compared to actual bodyweight unloading measured with scales [kg]
Number of device stops | Data are obtained during Appointment 1 between minute 25 and minute 45 and Appointment 2 between minute 10 to 30
  Number of Andago device stops measured throughout the habituation periods during appointments 1 and 2
Customized questionnaire investigating acceptability [dichotomous] | At the end of Appointments 1 (between minute 55-58) and the end of Appointment 2 (between minute 40-43)
  Participant is being asked whether the patient prefers treadmill or Andago (dichotomous outcome: 0=treadmill/1=Andago), and if the patient would like to train again in the Andago (0=no/1=yes). No sum score is calculated.
Questionnaire acceptability [visual analogue scale] | At the end of Appointments 1 (between minute 59-60) and the end of Appointment 2 (between minute 44-45)
  How much fun was it training in the Andago? [score 0=no fun at all to 10=maximal amount of fun]
Time needed for donning and doffing [seconds] | During Appointment 1 (mounting around minute 25; taking off around minute 43) and Appointment 2 (mounting around minute 1; taking off around minute 28)
  Time in seconds needed for mounting the patient in the Andago and, at the end of walking in the Andago, the time needed to get the patient out of the device
Manual Muscle Testing (MMT) | Appointment 1 between minute 1 and 5
  Manual muscle testing is performed for providing a characterization of the patients. For each muscle group, a score is given between 0 (no visible or palpable contraction) and 5 (patient moves over the full range of motion against gravity with additional maximal resistance). The following muscles will be tested: hip flexors and extensors; hip inner- and outer-rotators; knee flexors and extensors; ankle plantar and dorsal flexors
Selective Control Assessment of the Lower Extremity (SCALE) | Appointment 1 between minute 6 and 15 minutes
  The SCALE assesses the selectivity of lower extremity joints. It provides a score between 0 (not able) and 2 (normal selectivity) for each of the following joints: hip, knee, ankle, subtalar joint, and toes. It provides a sum score for the left and right leg separately (0= not able; 10= normal selectivity) and an overall sum score (0=not able; 20=normal selectivity)
Active and passive Range of Motion (ROM) of leg joints | Appointment 1 between minute 16 and 20 minutes
  Active (by patient) and passive (by therapist) mobility of the hip, knee and ankle joints are made in the sagittal plane. The ROM is noted according to the neutral zero method (degrees). ROM testing is performed for providing a characterization of the patients.
10 meter walk test | Appointments 1 between minute 21 and 25 and Appointment 3 between minute 1 and 5 and 56 and 60
  Children walk 14 meters; intermediate 10 meters is time stopped to calculate the walking speed

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Center of the University Children's Hospital, Affoltern am Albis, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
We have to check with the local ethics committee whether our pseudonymized data can be shared

REFERENCES:
- [Derived] van Hedel HJA, Rosselli I, Baumgartner-Ricklin S. Clinical utility of the over-ground bodyweight-supporting walking system Andago in children and youths with gait impairments. J Neuroeng Rehabil. 2021 Feb 8;18(1):29. doi: 10.1186/s12984-021-00827-1. PMID 33557834